CLINICAL TRIAL: NCT04508361
Title: Test-retest Reliability for Fatigue Assessment Scale, Short Form 6 Dimension and King's Sarcoidosis Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 248633
Record Dates: First submitted 2020-07-10; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to see if people's health related quality of life (how they feel about their health) changes over a 12 week period if they do not receive any change in their medicines. The investigators would like people to complete four questionnaires then repeat them after three months. The investigators need to do this to in order see what difference they should expect to detect if they give people treatment that works.

DETAILED DESCRIPTION:
Study Design This will be a questionnaire study, which will involve administering questionnaires to patients with sarcoidosis at baseline and after six and 12 weeks.

Participants can either complete the questionnaires whilst they are attending clinic, or alternatively return the questionnaires via a pre-paid postal envelope. The questionnaires will be administered at the same time; no other study measures will be taken subsequently. Demographic and clinical information will be collected from the patients' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged over 18
* Diagnosed with sarcoidosis by either; biopsy confirming non-caseating granulomas consistent with sarcoidosis, or multi-disciplinary interstitial lung disease meeting diagnosis of sarcoidosis
* Significant fatigue - defined as a FAS score of greater than 21 points
* Has mental capacity to complete the questionnaires

Exclusion Criteria:

* Presence of another significant cardio-respiratory disease, major organ disease (except where related to sarcoidosis) or chronic inflammatory condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with sarcoidosis and fatigue
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Assessment Scale (FAS) | Change from baseline to 12 weeks
  Fatigue Assessment Scale (FAS) - ranges from 10 to 50 with higher values representing greater fatigue. There are a specified cut-off values for clinically significant fatigue (score >= 22) and severe fatigue (score >= 35).The questionaire was administered at baseline, 6 weeks and 12 weeks.

SECONDARY OUTCOMES:
Short Form 36 (SF-36) | Change from baseline to 12 weeks
  Short Form 36 (SF-36) -ranges between 0 (maximum disability) and 100 (no disability). The SF36 score can be converted to utility scores using values within the questionnaire. The questionaire was administered at baseline, 6 weeks and 12 weeks.
Kings' Sarcoidosis Questionnaire (KSQ) | Change from baseline to 12 weeks
  Kings' Sarcoidosis Questionnaire (KSQ) ranges between 0 and 100 with higher numbers representing better health. The questionaire was administered at baseline, 6 weeks and 12 weeks.
Global rating of concept scale | Change from baseline to 12 weeks
  Global rating of concept scale. This is a ranking between 6 options to rate overall quality of life from no problem to very severe problem. The questionaire was administered at baseline, 6 weeks and 12 weeks.
The global rating of change | Change from 6 weeks to 12 weeks
  The global rating of change. This is a scoring out of 15 options to rate change in quality of life. It ranges between -7 and 7 with positive values representing an improvement. The questionaire was administered at 6 weeks and 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Norwich Medical School, Norwich, Norfolk, United Kingdom